CLINICAL TRIAL: NCT04327349
Title: Investigating Effect of Convalescent Plasma on COVID-19 Patients Outcome: A Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Shamshirian, Principal Investigator, Mazandaran University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR.MAZUMS.REC.1399.7330; IRCT20181104041551N1 (Registry Identifier: Iranian Registry of Clinical Trials (IRCT))
Record Dates: First submitted 2020-03-24; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Coronavirus Infections
Keywords: Coronavirus; COVID-19; SARS-CoV-2; Severe acute respiratory syndrome coronavirus 2
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 Patients (Other)
  Interventions: Biological: Convalescent Plasma

INTERVENTIONS:
Biological: Convalescent Plasma — Intervention to evaluate convalescent plasma transfer to COVID-19 patients admitted to ICU

SUMMARY:
Coronavirus disease 2019 (COVID-19) was recognized as a pandemic on March 11, 2020 by the World Health Organization. The virus that causes COVID-19 (SARS-CoV-2) is easily transmitted through person to person and there is still no specific approach against the disease and mortality rate in severe cases is also significant. Therefore, finding effective treatment for the mortality of these patients is very important. In this study the investigators aim to determine the effect of Convalescent Plasma on COVID-19 patients Outcome through a Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

Recipient:

1. COVID-19 Patients
2. Consent to attend the study
3. Age 30 to 70 years
4. Don't be intubated
5. PaO2 / FiO2 is above 200 or Spo2 is greater than 85%.

Donator:

1. Complete recovery from severe COVID-19 disease and hospital discharge
2. Consent to donate blood to the infected person
3. Age 30 to 60 years
4. Has normal CBC test results
5. Negative COVID-19 RT-PCR test

Exclusion Criteria:

Recipient:

1. A history of hypersensitivity to blood transfusions or its products
2. History of IgA deficiency
3. Heart failure or any other factor that prevents the transmission of of 500 ml plasma
4. Entering the intubation stage

Donator:

1. Patients infected with blood-borne viral / infectious diseases
2. Underlying heart disease, low or high blood pressure, diabetes, epilepsy, and anything that may prohibit blood donation.
3. Use of banned drugs for blood donation (eg, ethertinate, acitretin, aliotretinoin, isotretinoin, antiandrogens, NSAIDs, etc.)
4. Use of different drugs
5. Other prohibited donations based on blood transfusion standards

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-28 (Estimated); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Mortality changes in day 10 | 10 days after plasma transmission
  Measure of the number of deaths in a particular population, scaled to the size of that population, per unit of time.
Mortality changes in day 30 | 30 days after plasma transmission
  Measure of the number of deaths in a particular population, scaled to the size of that population, per unit of time.
Changes of C-reactive protein | Day 1
  Measurement of CRP
Changes of C-reactive protein | Day 3
  Measurement of CRP
Changes of C-reactive protein | Day 7
  Measurement of CRP
Changes of Interleukin 6 | Day 1
  Measurement of IL-6
Changes of Interleukin 6 | Day 3
  Measurement of IL-6
Changes of Interleukin 6 | Day 7
  Measurement of IL-6
Changes of tumor necrosis factor-α | Day 1
  Measurement of TNF-α
Changes of tumor necrosis factor-α | Day 3
  Measurement of TNF-α
Changes of tumor necrosis factor-α | Day 7
  Measurement of TNF-α
Changes of PaO2/FiO2 Ratio | Day 1
  Partial pressure of arterial oxygen/Percentage of inspired oxygen
Changes of PaO2/FiO2 Ratio | Day 3
  Partial pressure of arterial oxygen/Percentage of inspired oxygen
Changes of PaO2/FiO2 Ratio | Day 7
  Partial pressure of arterial oxygen/Percentage of inspired oxygen

SECONDARY OUTCOMES:
Changes of CD3 | Day 1
Changes of CD3 | Day 3
Changes of CD3 | Day 7
Changes of CD4 | Day 1
Changes of CD4 | Day 3
Changes of CD4 | Day 7
Changes of CD8 | Day 1
Changes of CD8 | Day 3
Changes of CD8 | Day 7
Changes of CD4/CD8 ratio | Day 1
Changes of CD4/CD8 ratio | Day 3
Changes of CD4/CD8 ratio | Day 7
Changes of lymphocyte count | Day 1
Changes of lymphocyte count | Day 3
Changes of lymphocyte count | Day 7
Changes of leukocyte count | Day 1
Changes of leukocyte count | Day 3
Changes of leukocyte count | Day 7
Changes of alanine transaminase (ALT) | Day 1
Changes of alanine transaminase (ALT) | Day 3
Changes of alanine transaminase (ALT) | Day 7
Changes of aspartate transaminase (AST) | Day 1
Changes of aspartate transaminase (AST) | Day 3
Changes of aspartate transaminase (AST) | Day 7
Changes of alkaline phosphatase (ALP) | Day 1
Changes of alkaline phosphatase (ALP) | Day 3
Changes of alkaline phosphatase (ALP) | Day 7
Changes of lactate dehydrogenase (LDH) | Day 1
Changes of lactate dehydrogenase (LDH) | Day 3
Changes of lactate dehydrogenase (LDH) | Day 7
Changes of creatine phosphokinase (CPK) | Day 1
Changes of creatine phosphokinase (CPK) | Day 3
Changes of creatine phosphokinase (CPK) | Day 7
Changes of Creatine kinase-MB (CK-MB) | Day 1
Changes of Creatine kinase-MB (CK-MB) | Day 3
Changes of Creatine kinase-MB (CK-MB) | Day 7
Changes of Specific IgG | Day 1
Changes of Specific IgG | Day 3
Changes of Specific IgG | Day 7
Radiological findings | Within 2 hours after admission
  Computed tomography Scan and Chest X-Ray
Radiological findings | Day 14
  Computed tomography Scan and Chest X-Ray
Number of days ventilated | Through study completion, an average of 2 weeks
Length of hospitalization | Through study completion, an average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Majid Saeedi, Ph.D., Study Chair — Vice-Chancellor for Research, Mazandaran University of Medical Sciences
Locations (1):
- Imam Khomeini Hospital, Mazandaran University of Medical Sciences, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: Undecided